CLINICAL TRIAL: NCT02817867
Title: Association Between Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation for Chronic Stroke Patients Rehabilitation: a Randomized Clinical Trial.
Brief Title: Association Between Brain Stimulations for the Rehabilitation of Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APPG-2016
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- tDCS (Active Comparator): Patients who will be treated with Transcranial direct-current stimulation (tDCS) in the ipsilesional motor cortex.
  Interventions: Device: tDCS
- rTMS (Active Comparator): Patients who will be treated with Magnetic brain stimulation (rTMS) in the contralesional motor cortex.
  Interventions: Device: TMS
- tDCS + rTMS (Experimental): Patients who will be treated with the association between Transcranial direct-current stimulation (tDCS) and magnetic brain stimulation (rTMS), in the ipsilesional and contralesional motor cortex, respectively.
  Interventions: Device: tDCS + TMS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation (tDCS)
  Arms: tDCS
Device: TMS — Transcranial magnetic stimulation
  Arms: rTMS
Device: tDCS + TMS — Association between tDCS and TMS.
  Arms: tDCS + rTMS

SUMMARY:
Cerebrovascular accident (CVA) is a cerebrovascular disease with high incidence and morbidity in the Brazilian population, and is considered a major cause of disability in adults. Brain damage caused by stroke generates a maladaptive pattern of neural activity and modulation between the cerebral hemispheres, unbalancing in the inter-hemispheric inhibition. This condition affects patient's functional recovery.

The aim of this study is to verify the effectiveness of repetitive transcranial magnetic stimulation Association (rTMS) in the cortex motor contralesional, Transcranial Direct Current Stimulation (tDCS) in the motor cortex ipsilesional and the association between these two types of brain stimulations on the upper limb recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subcortical stroke diagnosis, which has resulted in hemiparesis for at least 6 months and not more than 5 years (chronic condition);
* Ability to reach 60 degrees in the shoulder flexion
* Ability to completely extend the fingers in the affected upper limb;
* Minimal cognitive ability to understand commands;
* No current use of antiepileptic drugs for seizures.

Exclusion Criteria:

* Painful shoulder, adhesive capsulitis or glenohumeral subluxation;
* Contraindication (presence of metallic implants) or risks for the Transcranial magnetic stimulation, as evaluated by means of a standard questionnaire;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Motor Function by means of the Wolf Motor Function Test | change from pre to post (at least 10 days)

SECONDARY OUTCOMES:
Grip strength via hand dynamometer | change from pre to post (at least 10 days)
Manual Dexterity by means of the Box and Block Test | change from pre to post (at least 10 days)
Quality of Life by means of the Stroke Impact Scale | change from pre to post (at least 10 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil